CLINICAL TRIAL: NCT06155331
Title: Clinical Study to Evaluate the Possible Safety and Efficacy of Fenofibrate in the Prophylaxis of Doxorubicin Induced Cardiotoxicity in Breast Cancer Patients
Brief Title: Evaluation of Possible Safety and Efficacy of Fenofibrate in the Prophylaxis of Doxorubicin Induced Cardiotoxicity in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hagar Khaled Bassuony Dewidar, Instructor of clinical pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Breast cancer and fenofibrate
Record Dates: First submitted 2023-11-19; First posted 2023-12-04 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Stage 2 and 3
Keywords: Breast cancer , Doxorubicin, Fenofibrate , Cardiotoxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Fenofibrate; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): 22 patients which will receive four cycles of AC regimen (doxorubicin and cyclophosphamide; each cycle is given every 21 day) plus placebo tablets once daily.
  Interventions: Other: Placebo; Drug: Doxorubicin; Drug: Cyclophosphamide
- Fenofibrate group (Active Comparator): 22 patients which will receive four cycles of AC regimen (doxorubicin and cyclophosphamide; each cycle is given every 21 day) plus Fenofibrate 160 mg once daily.
  Interventions: Drug: Fenofibrate; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Fenofibrate — It is an approved drug for hypercholesterolemia, It lowers lipid levels by activating peroxisome proliferator-activated receptor alpha (PPARα).
  Arms: Fenofibrate group
Other: Placebo — Placebo is made to look exactly like a real drug but is made of an inactive substance.
  Arms: Placebo group
Drug: Doxorubicin — Anthracycline derived chemotherapy used in treatment of breast cancer
Drug: Cyclophosphamide — Alkylating agent used in treatment of breast cancer

SUMMARY:
This study aims at evaluating the possible safety and efficacy of fenofibrate in attenuating doxorubicin related cardiac toxicity in breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer represents the most frequently diagnosed malignancy and the second most common cause of cancer death worldwide (Sung et al., 2021). In Egypt, breast cancer is the most common malignancy in women, accounting for 38.8% of cancers in this population, with the estimated number of breast cancer cases nearly 22,700 in 2020 and forecasted to be approximately 46,000 in 2050 (Ibrahim et al., 2014).

Doxorubicin (DOX) is a cytotoxic agent that is commonly used for treatment of breast cancer. Despite its effectiveness, doxorubicin is associated with cumulative and potential cardiotoxicity (Rawat et al.,2021).

Although the precise mechanisms whereby DOX induces myocardial injury have not been fully elucidated, it is widely accepted that DOX induces cardiac injury via several mechanisms, including activation of nuclear factor- Kabba B (NF-ĸB), the induction of pro-inflammatory cytokines, the generation of free radicals, the promotion of apoptotic cell death, and the suppression of Endothelial progenitor cells (EPC) mobilization and function, which are typical changes observed in DOX-induced cardiotoxcity (Cardinale et al., 2020).

Peroxisome proliferator-activated receptor-α (PPARα) has been proposed as a key lipid metabolism modulator and regulator of inflammation. There are three isotypes of PPAR (α, β and ȣ) which have distinct but overlapping functions. Fenofibrate, an important PPAR- α agonist, is widely used in in the treatment for hypercholesterolemia and hypertriglyceridemia (Kim and Kim, 2020). Many studies demonstrated the pleiotropic effects of fenofibrate on the heart that afford direct myocardial protection in addition to the lipid-lowering effects through improvement of vascular endothelial function, reducing oxidative stress and increasing endothelial nitric oxide synthase (eNOS) activation (Walker et al., 2012; Jen et al., 2016).

In addition recent animal study showed that fenofibrate decreased the transactivation of Nuclear factor kappa-light-chain-enhancer of activated B cells (NF-κB), activated endothelial nitric oxide synthase (eNOS) and increased nitric oxide (NO) bioavailability, which in turn suppressed MMP-2 (matrix 4 metalloproteinase-2) and MMP-9 (matrix metalloproteinase-9), a well-recognized mediator of adverse ventricular fibrosis and subsequent remodeling, which established the role of fenofibrate against DOX-induced cardiotoxicity in mice (Huang et al., 2021). In addition, it is known that DOX- increases circulating N-terminal pro-B-type natriuretic peptide (NT- pro-BNP) and B-type natriuretic peptide (BNP) that were attenuated by fenofibrate (Huang et al., 2021)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients with biopsy confirmed diagnosis breast cancer and with stage II and stage III breast cancer according to the American Joint Committee on Cancer (TNM staging system of breast cancer).
* Patients with performance status <2 according to Eastern Cooperative Oncology Group (ECOG) score.
* Adequate baseline hematologic values (absolute neutrophilic count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L and hemoglobin level ≥ 10 g/dl).
* Patients with adequate liver function (serum bilirubin < 1.2 mg/dl) and adequate renal function (serum creatinine < 1.5 mg/d).

Exclusion Criteria:

* Patients with prior exposure to anthracyclines in the last 6 months.
* Patients with evidence of metastasis at the initial assessment.
* Concomitant use of antioxidant vitamins (vitamin A, C, E).
* Presence of clinical evidence for severe cardiac illness (angina pectoris, uncontrolled hypertension, arrhythmias and left ventricular ejection fraction <50%).
* Patients with inflammatory diseases (ulcerative colitis, rheumatoid arthritis).
* Patients with conditions associated with oxidative stress (smoking, tuberculosis, comorbid obesity).
* Patients who are candidates for monoclonal antibodies such as Trastuzumab and other targeted therapy (HER2 positive patients).
* Patients with active liver disease (cirrhosis, fatty liver, hepatitis C, etc..).
* Patients with myopathy.
* Patients with renal impairment, including those with end-stage renal disease and those receiving dialysis.
* Pregnant and breast feeding women.
* Known allergy to the fenofibrates.
* Concurrent use of statin, colchicine, ciprofibrate, idelalisib, ivacaftor, aspirin low strength, clopidogrel, warfarin, enzyme inducers (phenytoin, phenobarbitone, carbamazepine,…), enzyme inhibitors (allopurinol, MAOI, SSRI,…), drugs with high plasma protein binding capacity (sulfonamides, valproate, oral hypoglycemic, warfarin,…) in order to avoid potential pharmacodynamics and pharmacokinetic drug interactions.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in ejection fraction (the amount of blood that heart pumps each beat) using echocardiography | 3 months
  The primary outcome is to avoid decrease in patients ejection fraction while administrating doxorubicin which is known to cause a declination in cardiac ejection fraction threatening of heart failure

SECONDARY OUTCOMES:
Changes in serum levels of the measured biological markers | 3 months
  The secondary outcome is decrease in serum levels of the measured biological markers which are brain naturetic peptide and myeloperoxidase

CONTACTS AND LOCATIONS:
Overall Officials: Hagar Dewidar, Instructor, Principal Investigator — Tanta University
Locations (1):
- Hagar Dewidar, Tanta, Elgharbya, Egypt

REFERENCES:
- [Background] Amin MB, Greene FL, Edge SB, Compton CC, Gershenwald JE, Brookland RK, Meyer L, Gress DM, Byrd DR, Winchester DP. The Eighth Edition AJCC Cancer Staging Manual: Continuing to build a bridge from a population-based to a more "personalized" approach to cancer staging. CA Cancer J Clin. 2017 Mar;67(2):93-99. doi: 10.3322/caac.21388. Epub 2017 Jan 17. PMID 28094848
- [Background] Cardinale D, Iacopo F, Cipolla CM. Cardiotoxicity of Anthracyclines. Front Cardiovasc Med. 2020 Mar 18;7:26. doi: 10.3389/fcvm.2020.00026. eCollection 2020. PMID 32258060
- [Background] Czupryniak L, Joshi SR, Gogtay JA, Lopez M. Effect of micronized fenofibrate on microvascular complications of type 2 diabetes: a systematic review. Expert Opin Pharmacother. 2016 Aug;17(11):1463-73. doi: 10.1080/14656566.2016.1195811. Epub 2016 Jun 15. PMID 27267786
- [Background] Huang WP, Yin WH, Chen JS, Huang PH, Chen JW, Lin SJ. Fenofibrate attenuates doxorubicin-induced cardiac dysfunction in mice via activating the eNOS/EPC pathway. Sci Rep. 2021 Jan 13;11(1):1159. doi: 10.1038/s41598-021-80984-4. PMID 33441969
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] Jen HL, Liu PL, Chen YH, Yin WH, Chen JW, Lin SJ. Peroxisome Proliferator-Activated Receptor alpha Reduces Endothelin-1-Caused Cardiomyocyte Hypertrophy by Inhibiting Nuclear Factor-kappaB and Adiponectin. Mediators Inflamm. 2016;2016:5609121. doi: 10.1155/2016/5609121. Epub 2016 Oct 11. PMID 27807394
- [Background] Kim NH, Kim SG. Fibrates Revisited: Potential Role in Cardiovascular Risk Reduction. Diabetes Metab J. 2020 Apr;44(2):213-221. doi: 10.4093/dmj.2020.0001. PMID 32347023
- [Background] Rawat PS, Jaiswal A, Khurana A, Bhatti JS, Navik U. Doxorubicin-induced cardiotoxicity: An update on the molecular mechanism and novel therapeutic strategies for effective management. Biomed Pharmacother. 2021 Jul;139:111708. doi: 10.1016/j.biopha.2021.111708. Epub 2021 May 13. PMID 34243633
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Walker AE, Kaplon RE, Lucking SM, Russell-Nowlan MJ, Eckel RH, Seals DR. Fenofibrate improves vascular endothelial function by reducing oxidative stress while increasing endothelial nitric oxide synthase in healthy normolipidemic older adults. Hypertension. 2012 Dec;60(6):1517-23. doi: 10.1161/HYPERTENSIONAHA.112.203661. Epub 2012 Oct 29. PMID 23108655
- [Derived] Dewidar HK, Ghannam AA, Mostafa TM. Fenofibrate attenuates doxorubicin-induced cardiotoxicity in patients with breast cancer: a randomized controlled trial. Naunyn Schmiedebergs Arch Pharmacol. 2025 Dec;398(12):17109-17119. doi: 10.1007/s00210-025-04326-1. Epub 2025 Jun 3. PMID 40459761